CLINICAL TRIAL: NCT02585518
Title: Ecological Momentary Assessment of Eating Behavior in Overweight Youth
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Illinois Institute of Technology (Other); University of North Dakota (Other)
Responsible Party: Sponsor
Other Study IDs: IRB14-1212
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese: Children and adolescents with a BMI at or above the 85th percentile for age and sex
- Healthy control: Children and adolescents with a BMI below the 85th percentile for age and sex

SUMMARY:
The current study seeks to elucidate the context of pathological and non-pathological eating behavior in a heterogeneous sample of overweight and obese children, aged 8-14 years. Children will undergo a two-week ecological momentary assessment (EMA) protocol in which they record all eating episodes and their physiological, emotional, interpersonal, and environmental correlates. Specific aims are to identify proximal antecedents and consequences of pathological and non-pathological eating in overweight and obese children, and to determine the prevalence of loss of control eating in the natural environment.

DETAILED DESCRIPTION:
Interested individuals will be screened via phone for initial study eligibility. Potentially eligible participants and their parents will attend an in-person screening at the University of Chicago in which they will complete assent and consent procedures. Youth will have their height and weight measured and complete interviews to assess eating disorder symptoms and psychiatric comorbidities. Eligible participants and parents will then complete self- and parent-report assessments of eating behavior, body image concerns, psychiatric symptoms, and interpersonal functioning. Participants will then be trained on how to complete the EMA recordings.

A one-day practice period during which adherence is ≥70% of ratings will qualify children to initiate the 14-day EMA study period; these data will not be used in statistical analyses to reduce concerns about the effect of immediate reactivity to self-monitoring. Youth will self-monitor on a smartphone or other wireless device through the use of the ReTAINE (Real-Time Assessment in the Natural Environment) system. ReTAINE™ is a secure, web-based system that allows for momentary data to be collected through a wide variety of portable devices. Youth may use their own smartphone/wireless device or one provided by the study team. Recent survey data suggest that up to 80% of children and adolescents have access to the Internet through a cellular phone or other wireless device, indicating that this approach is reasonable in this age group. EMA protocols have been completed with good compliance in youth.

The proposed study will include three types of EMA signaling methods.63 First, participants will be signaled at 3-5 semi-random times throughout the day (signal-contingent) to report on current affect, stressors, interpersonal functioning, and to report any eating episode that has not been previously recorded. These signals will occur at random times between 7:00-8:00am, 3:00-4:00pm, and 6:00-7:00pm on weekdays, so as not to interfere with the school day; and between 8:00-9:00am, 11:00am-12:00pm, 2:00-3:00pm, 5:00-6:00pm, and 8:00-9:00pm on weekend days. In addition, participants will be instructed to complete momentary ratings of affect, stressors, interpersonal functioning, and a variety of physiological, environmental, cognitive, and behavioral factors associated with eating as soon after each eating episode as possible (event-contingent). Event-contingent ratings will allow for the assessment of immediate consequences of eating that may be missed by the random signals. Finally, participants will complete ratings of affect, stressors, interpersonal functioning, and physiological, environmental, cognitive, and behavioral factors at the end of each day (interval-contingent) to capture any changes since the last random signal. This combination of signal-, event-, and interval- contingent recordings has been successfully implemented in previous EMA studies of overweight youth.

Participants will be contacted by phone after the first day of EMA recording, at which point they will be given feedback regarding their compliance rates, and any questions or concerns regarding assessment procedures will be discussed with a research assistant. Throughout the 14-day assessment period, we will also attempt to contact participants via telephone at least twice per week to check in with them regarding any problems or concerns. This approach has demonstrated success in participant retention and validated compliance during a previous research study which required daily collection of saliva samples and interval ratings of mood and disordered eating behaviors over 35 days.

Complementary to the collection of EMA data, Nutritional Data System for Research (NDS-R)65 will be used to compile nutritional intake data on eating episodes reported by participants through the ReTAINE system. Two weekdays and one weekend day during the 14-day protocol will be randomly selected for each participant, during which the participant will be contacted by phone and asked to recall the details of each of that day's eating episodes. The time points of each eating episode will be entered into the NDS-R system, and the nutritional data of interest will be merged with the EMA data in order to assess contextual factors associated with specific dietary patterns (e.g., consumption of high fat meals). ActiGraph watches (GT3X) will be worn by participants for the duration of the 14-day protocol to compile data on sleep patterns in the natural home environment. These computerized wristwatch-like devices collect data generated by movement and are minimally invasive. Participants' parents will also complete 14-day sleep diaries in which they will record their children's bedtime and wake time, which will provide the start and end times for actigraphy analyses.

At the completion of the daily assessment phase, participants will return to the University of Chicago to return the loaner smartphone, if applicable; complete a brief, final assessment; and receive their final study incentive payments. The final assessment will include a modified version of the Child Eating Disorder Examination (ChEDE) interview to cover the previous two weeks during which EMA was conducted. This assessment will be used to determine changes in symptom frequency (i.e., reactivity to study procedures).

ELIGIBILITY:
Inclusion Criteria:

Participants be included if they are overweight or obese (BMI≥85th %ile) and aged 8-14 years.

Exclusion Criteria:

Participants will be excluded if they 1) are currently taking any medications known to affect weight or appetite (e.g., antidepressants, steroids, chemotherapy drugs); 2) have a current or past diagnosis of an eating disorder involving purging or suppressed body weight (e.g., bulimia nervosa or anorexia nervosa); 3) are unable to read and understand English fluently; or 4) are receiving concurrent treatment for obesity.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will comprise 40 overweight or obese (BMI≥85th %ile) youth aged 8-14 years. Every effort will be made to recruit a racially/ethnically diverse sample. Participants will be excluded if they 1) are currently taking any medications known to affect weight or appetite (e.g., antidepressants, steroids, chemotherapy drugs); 2) have a current or past diagnosis of an eating disorder involving purging or suppressed body weight (e.g., bulimia nervosa or anorexia nervosa); 3) are unable to read and understand English fluently; or 4) are receiving concurrent treatment for obesity.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-02; Primary Completion 2017-01-21 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Eating episodes | Repeated measures throughout the 2-week EMA protocol

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Goldschmidt, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States